CLINICAL TRIAL: NCT04277078
Title: Predicting Factors of Intubation in Hospitalised Patients With Acutely Attacked Asthma
Brief Title: Predicting Intubation of Patients Hospitalised for Acutely Attacked Asthma
Status: Completed | Type: Observational
Sponsor: Hat Yai Medical Education Center (Other)
Responsible Party: Principal Investigator, Narongwit Nakwan, Asst.prof, Hat Yai Medical Education Center
Other Study IDs: 65/2562
Record Dates: First submitted 2020-02-15; First posted 2020-02-20 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2020-02

CONDITIONS: Intubation Complication; Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intubated asthma attack: Patients who had been hospitalised with asthma attack, then intubated during hospitalisation.
- Non-Intubated asthma attack: Patients who had been hospitalised with asthma attack without intubation during hospitalisation.

SUMMARY:
Although the asthmatic treatments currently be effective in term of efficacy of inhaled medications and good clinical outcome including symptom controlled and asthma exacerbation number, the large number of worse event still have been reported. Few cases eventually have been intubated and died even though using optimal medication. In this study, we will search to identify factors that may influence intubation in hospitalised patient with asthmatic attack.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had been admitted and diagnosed as asthmatic attack between year 2016-2018.
* Patients who have age > 15 year old.

Exclusion Criteria:

* Non

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Population in this study is a the patient who had been admitted with moderate to severe asthmatic attack. The study will be retrospective review with data in medical record between year 2016-2018. The baseline characteristic and factors which has a potential to intubation will be recored.
Sampling Method: Non-Probability Sample
Enrollment: 509 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
Number case of intubated patient | Retropectively review 2 years backard between 2017-2018
  Number case of hospitalized asthmatic attack patients during 2-year review.

SECONDARY OUTCOMES:
Number of previous asthma attack before this admission | 1 year before admission
  Number of previous asthma attack with 12 months before this hospitalization.
Blood eosinophil count at admission time | Retropectively review 2 years backard between 2017-2018
  Blood eosinophil may help predict outcome and risk for intubation.
Number patients dead | Retropectively review 2 years backard between 2017-2018
  Number patient dead during hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Narongwit Nakwan, M.D., Principal Investigator — HatYai Hospital
Locations (1):
- Hatyai Hospital, Hat Yai, Changwat Songkhla, Thailand

IPD SHARING:
Plan to Share IPD: No